CLINICAL TRIAL: NCT06613191
Title: P2Y12 Inhibitor Versus Aspirin Monotherapy in Patients Undergoing Elective Screening and Surveillance Colonoscopy
Brief Title: Colonoscopy and Antiplatelet Therapy Trial
Acronym: CAPTT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ochsner Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2024.105; INVEST CVD (Other: Ochsner Clinic Foundation)
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Coronary Arterial Disease (CAD); Peripheral Vascular Disease
Keywords: Colonoscopy; Antiplatelet therapy
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Aspirin; Clopidogrel; Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin only (Active Comparator): Participants receiving aspirin only at time of the colonoscopy
  Interventions: Drug: Aspirin
- P2Y12 inhibitor only (Experimental): Participants receiving a P2Y12 inhibitor only at time of the colonoscopy
  Interventions: Drug: P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel)

INTERVENTIONS:
Drug: Aspirin — Participant will be on aspirin alone or P2Y12 inhibitor alone
  Arms: Aspirin only
Drug: P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel) — Participant will be taking either P2Y12 inhibitor at time of colonoscopy
  Arms: P2Y12 inhibitor only

SUMMARY:
Patients on dual antiplatelet therapy )aspirin plus a P2Y12 inhibitor [clopidogrel, prasugrel, or ticagrelor]) undergoing screening or surveilance colonoscopy are at increased risk for bleeding from the procedure. Patients are ussually asked to stop the P2Y12 inhibitor for the procedure. Currently, recommendation is that patients only on a P2Y12 inhibitor be changes to aspirin for the procedure. This pilot study will evaluate if there is a large difference in bleeding between patients only taking aspirin compared with patients only taking a P2Y12 inhibitor. Patinets who participate will randomly be randomly asked to stop either aspirin or the P2Y12 inhibitor 1 week before the procedure. Periprocedural bleeding and bleeding after the procedure for iup to 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 45 years
2. Stable patients defined as having Angina CCS (Canadian Cardiovascular Society) class 1-3 and/or Heart Failure NYHA class 1-2 without a change in guideline directed anti-ischemic or heart failure medications within 30 days prior to randomization.
3. Patients with cardiovascular disease defined as coronary artery disease, cerebrovascular disease or peripheral vascular disease taking DAPT (defined as aspirin plus a P2Y12 inhibitor). The decision to use DAPT in this patient will be made by the managing physician(s) before recruitment for this study. Consider replacing last statement with "As directed by their physician prior to recruitment into this study"
4. Scheduled for elective screening or surveillance outpatient colonoscopy

Exclusion Criteria:

1. Coronary intervention (PCI or CABG) less than 90 days prior to randomization
2. ACS event in less than 90 days prior to randomization
3. Transient ischemic attack (TIA) and/or stroke event in less than 90 days prior to randomization
4. Acute limb ischemia and/or amputation in less than 90 days prior to randomization
5. Post cardiac valve replacement (either percutaneous or surgical)
6. High cardiovascular risk:

   1. Patients with CCS class 4 angina
   2. Hospitalized with ACS within 1 month prior to randomization
   3. Patients undergoing PCI or CABG within the 3 months prior to randomization
7. Patients on left ventricular assist device (LVAD) or post cardiac transplantation
8. Patients with NYHA class 3 or 4 heart failure
9. Any condition requiring treatment requires chronic use of an anticoagulant.
10. Chronic kidney disease Stage 5 (with or without dialysis)
11. Liver cirrhosis with platelet count < 50,000/ mm3 and/or INR >1.4
12. Hematocrit < 30% and hemoglobin < 10 mg/dL
13. Emergent or inpatient Colonoscopy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpont | 7 days
  Composite of:
  * Use of endoscopic clips post-polypectomy to control persistent intraprocedural bleeding (defined as bleeding persisting for greater than 2 minutes),
  * Major delayed bleeding, which was symptomatically or clinically overt and associated with an unplanned admission or readmission to hospital for rectal bleeding,
  * Bleeding that directly contributed to death,
  * Minor bleeding defined as any sign or symptom of peri-rectal bleeding that did not fit the above criteria,
  * Need for further intervention to control bleeding such as endoscopic, surgical, or radiological intervention, or
  * Bleeding causes a fall in hemoglobin ≥ 2 g/dL or leads to transfusion of whole blood or red cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Ochsner Health, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided